CLINICAL TRIAL: NCT00148252
Title: Lowering Total Immunosuppressive Load in Renal Transplant Recipients More Than 12 Months Posttransplant - Randomised Withdrawal of Mycophenolate Mofetil (CellCept®) or Cyclosporine A (Sandimmun Neoral®)
Brief Title: Lowering Total Immunosuppressive Load in Renal Transplant Recipients More Than 12 Months Posttransplant
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: To high rejection rate in CsA withdrawal arm
Sponsor: University of Oslo School of Pharmacy (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NILS 02-08144
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Renal Transplantation
Keywords: Calcineurin; reduction; immunosuppression; cyclosporine A; mycophenolate mofetil

INTERVENTIONS:
Drug: Mycophenolate mofetil withdrawal
Drug: Cyclosporione A withdrawal

SUMMARY:
To compare the change in renal function between CsA or MMF withdrawal from before to 12 months after drug withdrawal in renal transplant recipients on triple immunosuppressive therapy

DETAILED DESCRIPTION:
To compare the change in renal function between CsA or MMF withdrawal from before to 12 months after drug withdrawal in renal transplant recipients on triple immunosuppressive therapy.

Secondly to examine safety following withdrawal of CsA or MMF, respectively, by the following parameters:

* Biopsy verified acute rejection episodes, time to first rejection and number of steroid resistant rejection episodes within 12 months.
* Hematology (Hb, WBC, platelets) abnormalities within 12 months.
* Graft and patient survival at 12 months and 5 years. Absolute difference in renal function between withdrawal groups at 12 months. Three monthly changes in renal function from drug withdrawal to 12 months. Change in dyslipidemia frequency from drug withdrawal to 12 months. Change in hypertension frequency from drug withdrawal to 12 months. Change in glucose tolerance from drug withdrawal to 12 months. Cumulative incidence of clinical infections resulting in hospitalization within 12 months.

Sub protocols will also examine the following aspects:

Cardiovascular: Homocysteine. Lipid peroxidation. Microvascular function and vasoactive parameters Quality of life (QoL): ESRD SCL-TM, SF-36 (short version) and EQ-5D (GI-checklist extended) questionnaires will be used.

Pharmacoeconomical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients of either gender above 18 years of age at time of randomisation. 2. More than twelve months posttransplant. 3. Treated with an immunosuppressive protocol consisting of CsA, MMF and steroid from the time of discharge from the transplant clinic (e.g. 3 months posttransplant).

  4. Kidney (only) transplant recipients with stable renal function (S-creatinine < 300 umol/L and an average increase in S-creatinine < 20% the last 6 months prior to inclusion) and without treated clinically and/or biopsy proven acute rejection episodes the last 6 months prior to inclusion.

  5. No previous steroid resistant acute rejections (e.g. treated with ATG/OKT3). 6. Not more than two steroid sensitive acute rejections posttransplant. 7. Signed informed consent.

Exclusion Criteria:

- 1. PRA positivity > 20%. 2. Concomitant therapy with other investigational drugs or prohibited medication specified in the protocol.

3. Life expectancy less than one year. 4. Acute illness or acute fungal, bacterial or viral infection at screening. 5. Unable and/or unlikely to follow the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298
Dates: Start 2003-02; Primary Completion 2005-11 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the absolute change in renal function from inclusion to 12 months post drug withdrawal, evaluated as GFR estimated from Nankivell's formula B and normalised for 1.73 m2 body-surface.

SECONDARY OUTCOMES:
Graft and patient survival at 12 months and 5 years posttransplant.
Proportion of patients with biopsy-proven acute rejection or acute rejection (biopsy proven + presumptive) episodes within 12 months.
Incidence of HB, WBC, platelet abnormal values requiring clinical intervention within 12 months.
Incidence of need for additional immunosuppressive therapy at 12 months.
Absolute difference in renal function between treatment groups at 12 months, evaluated by Nankivell's formula (B).
Renal function (Nankivell's formula B) development over time (3 monthly) between treatment groups within 12 months.
Change in dyslipidemia frequency from drug withdrawal to 12 months.
Change in hypertension frequency from drug withdrawal to 12 months.
Change in glucose tolerance from drug withdrawal to 12 months.
Cumulative incidence of clinical infections resulting in hospitalization within 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Åsberg, MSc, Study Director — University of Oslo
Locations (9):
- Norway (9):
  - Rikshospitalet, Section of Nephrology, Oslo, Oslo County
  - Haukeland sykehus, Bergen
  - Lillehammer hospital, Lillehammer
  - Akershus Hospital, Nordbyhagen
  - Ullevål hospital, Oslo
  - Hospital Telemark, Skien
  - Sentralsykehuset i Rogaland, Stavanger
  - Tromsø hospital, Tromsø
  - St. Olavs hospital, Trondheim

REFERENCES:
- [Derived] Asberg A, Apeland T, Reisaeter AV, Foss A, Leivestad T, Heldal K, Thorud LO, Eriksen BO, Hartmann A; NILS Study Group. Long-term outcomes after cyclosporine or mycophenolate withdrawal in kidney transplantation - results from an aborted trial. Clin Transplant. 2013 Mar-Apr;27(2):E151-6. doi: 10.1111/ctr.12076. Epub 2013 Jan 27. PMID 23351013